CLINICAL TRIAL: NCT02019134
Title: A Randomized Pragmatic Trial About the Effectiveness of an App Based Relaxation Technique for Patients With Chronic Neck Pain
Brief Title: Effectiveness of App-based Relaxation for Patients With Chronic Neck Pain
Acronym: Relaxneck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof Dr. Claudia M. Witt, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Relaxneck-13
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Chronic Neck Pain
Keywords: chronic neck pain; relaxation technique; comparative effectiveness research
MeSH Terms: interventions — Meditation; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care waiting list (Active Comparator): Patients allocated to the usual care waiting list group will continue with their usual care without receiving any additional therapy
  Interventions: Other: ususal care
- relaxation exercise (Experimental): Participants allocated to the relaxation group will apply daily but at least five days a week a 15-minutes relaxation exercise, guided by a smartphone application (App). On a daily basis, participants can select one out of the three exercises (guided imagery, mindfulness based training, autogenic training) which they want to apply
  Interventions: Behavioral: relaxation exercise

INTERVENTIONS:
Behavioral: relaxation exercise — relaxation exercise
  Other Names: meditation
  Arms: relaxation exercise
Other: ususal care
  Other Names: waiting list
  Arms: usual care waiting list

SUMMARY:
The aim of the pragmatic randomized study is to evaluate whether additional relaxation technique is more effective in the reduction of chronic neck pain compared to usual care alone.

DETAILED DESCRIPTION:
Objective: To evaluate whether additional relaxation technique is more effective in the reduction of chronic neck pain compared to usual care alone.

Study design: Open single-centered randomized two-armed pragmatic trial.

Participants: 220 patients aged 18-65 years with chronic (>12 weeks) neck pain and a mean pain score ≥ 4 on a Numeric Rating scale (NRS) in the last week before randomization who will be randomly allocated to two groups (relaxation, usual care alone as waiting list)

Intervention: Participants apply either a daily 15-minute relaxation exercise guided by a smartphone application ("app"). or apply no additional intervention. The exercise should be applied daily, (minimally, five days per week) for 6 months. The app contains audios to guide autogenic training, muscle relaxation training and guided imagery. On a daily basis, participants can select one of the three exercises which they want to apply.

Main outcome measure: The primary outcome is the mean pain intensity after 3 months measured by the daily pain intensity on the NRS.

ELIGIBILITY:
Inclusion Criteria:

* female or male
* 18-65 years of age
* chronic neck pain for at least 12 weeks
* if additional back pain is reported, neck pain has to be predominant
* intensity of the average neck pain ≥ 4 on the numeric rating scale (NRS) in the last week
* presence of a smartphone (iphone, Android phone) and willingness to do data entry through a smart phone application (App)
* physical and mental ability to participate in the study
* willingness to be randomized, to apply study intervention according to the protocol, to complete the baseline questionnaire in paper form and electronic questionnaires and diaries provided by a smart phone application
* written and oral informed consent

Exclusion Criteria:

* neck pain caused by a known malignant disease
* neck pain caused by trauma
* known rheumatic disorder
* history or planned surgery of the spinal column of the neck in the next 6 months
* known neurological symptoms e.g radicular symptoms because of prolapsed vertebral disc
* regular intake of analgesics (>1x per week) because of additional diseases
* intake of centrally acting analgesics
* known severe acute or chronic disorder, that do not allow participation in the therapy
* other known diseases, that do not allow participation in the therapy
* known alcohol or substance abuse
* no sufficient German language skills
* current application for a benefit
* participation in another clinical trial during six months before the study and parallel to the study
* conducting regular relaxation techniques, mindfulness training or meditation six weeks before the study or planned in the next 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Primary outcome is the mean pain intensity over 3 months measured by the daily pain intensity on the Numeric rating scale (NRS) | 3 months

SECONDARY OUTCOMES:
Mean pain intensity measured by the daily pain intensity on the NRS | 6 months
Mean pain intensity measured weekly as the average pain intensity of the last seven days on a NRS | 3 and 6 months
Pain acceptance | 3 and 6 months
  German version of Chronic Pain Acceptance Questionnaire
Stress | 3 and 6 months
  NRS
Suspected adverse reaction | 3 and 6 month
Number of serious adverse event | 3 and 6 month
medication intake | 3 and 6 months
Number of sick leave days | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, Prof. Dr. med, Principal Investigator — Institute for Social Medicine, Epidemiology and Health Economics, Charité - Universitätsmedizin Berlin
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Pach D, Blodt S, Wang J, Keller T, Bergmann B, Rogge AA, Barth J, Icke K, Roll S, Witt CM. App-Based Relaxation Exercises for Patients With Chronic Neck Pain: Pragmatic Randomized Trial. JMIR Mhealth Uhealth. 2022 Jan 7;10(1):e31482. doi: 10.2196/31482. PMID 34994708
- [Derived] Blodt S, Pach D, Roll S, Witt CM. Effectiveness of app-based relaxation for patients with chronic low back pain (Relaxback) and chronic neck pain (Relaxneck): study protocol for two randomized pragmatic trials. Trials. 2014 Dec 15;15:490. doi: 10.1186/1745-6215-15-490. PMID 25511185